CLINICAL TRIAL: NCT05908604
Title: The Effect of a Robot in Medication Management for Older People's Home Care: a Non-randomized Controlled Clinical Trial
Brief Title: Use of a Robot in Medication Management for Older People's Home Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Savonia University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Riitta Turjamaa, Post doc researcher, Director of Continuous Learning, Savonia University of Applied Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: University of Eastern Finland
Record Dates: First submitted 2023-05-06; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Unrecognized Condition
Keywords: home-care professional; medication management; older people's home care; robot; working time

STUDY DESIGN:
Intervention Model Description: Non-randomized controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): In the IG, home care professionals load medications inside the robot, and it enabled older home care clients to carry out medication management by themselves.
  Interventions: Other: Robot for madication management
- Control group (Sham Comparator): In the CG, home care professionals manually dispensed medications to doset and administrating medications during their home visits.
  Interventions: Other: Robot for madication management

INTERVENTIONS:
Other: Robot for madication management — The effect of a robot in medication management for older people's home care

SUMMARY:
Non-randomized controlled clinical trial was used. Data were collected using the Working Time Tracking Form in three data collection points (baseline, at 1 month and at 2 month). The participants were home care professionals who carried out home care clients' medication management. Home care clients were allocated into intervention and control groups (n=64 and 46, respectively) based on whether or not they used the robot. The statistical analysis methods were used.

DETAILED DESCRIPTION:
The data were collected using a Working Time Tracking Form, which was developed by professional team for this study. The team included senior lecturer in nursing with medication management competence, head of older people's home care, and home care professional working in older people's home care. The content of the Time Tracking Form was founded on previous literature about the medication management process in home care. The research protocol was planned by the authors before the study and it can be accessed from the corresponding authors on a reasonable request. The home care professionals filled in the Working Time Tracking Form the time in minutes they used for each phase of process i.e. ordering medications, dispensing medications to the doset or dispensing medications to the robot, reconstitution medications, administration of medications in tablets, administration of medications in other routes, medication education, and monitoring the effects of medications. The Working Time Tracking Form was filled in from each client and from each home visit, which included medication management for a five-day period in baseline and in follow up after one and two months.

The expert panel evaluated, and pilot group pre-tested the Time Tracking Form's content validity. The expert panel consisted of seven participants: one head of home care, three home care professionals, and two senior lecturers in nursing with medication management competence, and one statistician. Panel members evaluated each item focusing on usability, but they did not find revision. A pre-test (answers were not included in this study) was performed with 10 home care professionals having the experience using the robot for medication management in older people's home care. This helped evaluate how understandable and clear the Time Tracking Form's content was and how long time it took to be completed.

The SPSS v.26 software was used to analyse data.The characteristics of sample were reported using descriptive statistics including frequencies, percentages, medians, mean values, and standard deviation.

ELIGIBILITY:
Inclusion Criteria:

* voluntariness,
* working presently in older people's home care and
* communication in Finnish or English

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Baseline measurement: working time used for medication management during one week | One week
  Data were collected using the Working Time Tracking Form. The participants were home care professionals who carried out home care clients' medication management. Home care clients were allocated into intervention and control groups (n=64 and 46, respectively) based on whether or not they used the robot. The statistical analysis methods were used.
Change from baseline working time used for medication management at 1 month during one week | One week
  Data were collected using the Working Time Tracking Form. The participants were home care professionals who carried out home care clients' medication management. Home care clients were allocated into intervention and control groups (n=64 and 46, respectively) based on whether or not they used the robot. 1-month measurement was carried out one month after the baseline measurement. The aim of the measurement was to evaluate the change of using a robot for medication management on home care professionals' use of working time.
Change from baseline working time used for medication management at 2 months during one week | One week
  Data were collected using the Working Time Tracking Form. The participants were home care professionals who carried out home care clients' medication management. Home care clients were allocated into intervention and control groups (n=64 and 46, respectively) based on whether or not they used the robot. 2-month measurement was carried out two month after the baseline measurement. The aim of the measurement was to evaluate the change of using a robot for medication management on home care professionals' use of working time.

CONTACTS AND LOCATIONS:
Overall Officials: Riitta Turjamaa, PhD, Principal Investigator — Savonia University of Applied Sciences
Locations (1):
- Riitta Turjamaa, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kajander-Unkuri S, Vaismoradi M, Katajisto J, Kangasniemi M, Turjamaa R. Effect of robot for medication management on home care professionals' use of working time in older people's home care: a non-randomized controlled clinical trial. BMC Health Serv Res. 2023 Dec 2;23(1):1344. doi: 10.1186/s12913-023-10367-0. PMID 38042773